CLINICAL TRIAL: NCT02533219
Title: Phase II Study of the Use of [18F]-DOPA in Hyperinsulinemic Hypoglycemia
Brief Title: Study of the Use of [18F]-DOPA in Hyperinsulinemic Hypoglycemia
Acronym: [18F]-DOPA
Status: No longer available | Type: Expanded Access
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Victor J. Seghers, Assistant Professor of Radiology, Baylor College of Medicine
Other Study IDs: H-32432
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Hyperinsulinemic Hypoglycemia, Persistent; Congenital Hyperinsulinism; Persistent Hyperinsulinemic Hypoglycemia of Infancy (PHHI)
Keywords: Hyperinsulinemic hypoglycemia; PET/CT; PET/MRI; [18F]-DOPA; PET/MR; Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — fluorodopa F 18

INTERVENTIONS:
Drug: 18 F-DOPA — Subjects will undergo PET imaging with [18F]-DOPA. All PET imaging will be performed after administration of a single dose (0.08 - 0.16 mCurie/kg) of [18F]-DOPA. PET imaging can be performed on either Philips Ingenuity TF PET/MRI or PET/CT.
  Other Names: Fluorine-18-L-dihydroxyphenylalanine

SUMMARY:
The primary objective of this study is to evaluate the utility of [18F]-DOPA PET to provide improved presurgical planning and distinguish between focal and diffuse forms of HI. The investigators will perform descriptive analysis, relying on visual analysis to diagnose and localize a focal lesion. Our findings will be compared to surgical histopathology to determine sensitivity and specificity or this technique. The investigators will also track patient surgical outcomes, specifically whether the patient is surgically "cured" or still requires medical management to control residual hypoglycemia.

DETAILED DESCRIPTION:
Hyperinsulinemic hypoglycemia is caused by low glucose due to excessive insulin secretion and remains difficult to treat because of the requirement for extensive amounts of glucose and the lack of effective long-term medical therapy. Correct diagnosis, localization, and limited excision of the focal lesion will result in a complete cure of the patient. In contrast, medically unresponsive diffuse disease requires a near total pancreatectomy, greatly increasing the risk of future diabetes mellitus. Fortunately, [18F]-DOPA PET has been shown to be a useful noninvasive imaging method for distinguishing between focal and diffuse forms of hyperinsulinemic hypoglycemia. In this study, the investigators seek to validate the effectiveness of using PET/MR and PET/CT with F-DOPA to accurately and reliably detect and localize disease.

ELIGIBILITY:
Inclusion Criteria:

* All Patients clinically diagnosed with Hyperinsulinemia of any age
* Patients in need of PET scan
* Patients that require sedation
* Patients that do not require sedation

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Patients without Hyperinsulinemia
* Patients who are or may be pregnant
* Serious intercurrent medical illness other than hypoglycemia that precludes having the scan either because of patient instability or concerns about potential toxicity.
* Patient's requiring emergency surgical intervention that would be inappropriately delayed by [18F]-DOPA PET imaging.

Max Age: 64 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States